CLINICAL TRIAL: NCT03272412
Title: Impact of Serum Progesterone Levels on the Day of Embryo Transfer in Artificial Endometrial Preparation Cycles on the Ongoing Pregnancy Rate.
Brief Title: Serum Progesterone on the Day of Embryo Transfer and Pregnancy Rate.
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Elena Labarta, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 1704-VLC-024-EL
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ongoing Pregnancy Rate
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Analysis of serum Progesterone in blood sample — Levels of progesterone will be determined on the day of embryo transfer in patients undergoing artificial endometrial preparation cycles.

SUMMARY:
This study aims to analyze whether serum Progsterone levels on the day of Embryo Transfer are related with Ongoing Pregnancy rate in artificial endometrial preparation cycles with intravaginal micronized progesterone.

ELIGIBILITY:
Inclusion Criteria

1. Age <50 years old
2. Hormonal Replacement therapy cycle for embryo transfer in any of the following situations:

   1. Embryos in fresh cycle with donated oocytes.
   2. Subsequent embryo transfers of vitrified embryos in cycles of donated oocytes.
   3. Frozen embryo transfers in cycles with autologous oocytes.
3. Endometrial line: >6.5-7mm (with trilaminar aspect) in proliferative phase, before introducing progesterone.
4. Administration of natural micronized progesterone intravaginally (400 mg/12 hours for 5 complete days (10 dosis), before the embryo transfer and maintained until pregnancy week 12.
5. Embryo transfer of blastocyst (day 5-6).
6. Signed Informed Consent

Exclusion Criteria

1. Uterine pathology (submucous o intramural fibroids (>4 cm) or which deform the uterine cavity; endometrial polyps or Müllerian anomalies; or adnexal anomalies (communicating hydrosalpinx).
2. Simultaneous participation in another clinical study.
3. Participation in another clinical study before the inclusion in the present study, and which could affect the objectives of the present study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women who are undergoing IVF treatments with artificial endometrial preparation with hormonal replacement therapy.
Sampling Method: Probability Sample
Enrollment: 1205 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Concentration of serum Progesterone levels | The day of embryo transfer
  Serum progesterone levels
Ongoing Pregnancies depending on Progesterone levels ranges. | Week 5-12 after Embryo Transfer
  Ultrasound to confirm Ongoing Pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Spain

REFERENCES:
- [Derived] Labarta E, Mariani G, Paolelli S, Rodriguez-Varela C, Vidal C, Giles J, Bellver J, Cruz F, Marzal A, Celada P, Olmo I, Alama P, Remohi J, Bosch E. Impact of low serum progesterone levels on the day of embryo transfer on pregnancy outcome: a prospective cohort study in artificial cycles with vaginal progesterone. Hum Reprod. 2021 Feb 18;36(3):683-692. doi: 10.1093/humrep/deaa322. PMID 33340402